CLINICAL TRIAL: NCT04230005
Title: How is it to Work With JEMS: Physiotherapists' Experiences in Working With Joanne Elphinston Movement Systems, JEMS, in Primary Care Rehabilitation A Focusgroup Study
Brief Title: How is it to Work With JEMS: Physiotherapists' Experiences in Working With JEMS, in Primary Care Rehabilitation
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 270851
Record Dates: First submitted 2020-01-12; First posted 2020-01-18 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-06

CONDITIONS: Injuries
Keywords: Movement; Rehabilitation; Learning
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In Physiotherapy movement is a central concept and a clinical tool. Different methods are developped for analysing and assessing movement patterns offering patients a more functional way in moving and enable performance development i daily activities and sports.

The aim of this focusgroup study is to illustrate physiotherapists' experiences using the method JEMS working with patients in rehabilitation in Primary Care.

Possible benefits of the study: There is a need for in-depth knowledge of colleagues' experiences and experiences about what it is like using the JEMS concept in the clinic. The results can be used as a discussion basis in a counseling context, be developmental for the individual physiotherapist and a guidance when different methods for movement analysis and treatment / training are to be chosen when implementing in clinical rehabilitation activities.

DETAILED DESCRIPTION:
The physiotherapist works with movement as a main mean of promoting health and reducing illness. At disposal, the physiotherapist has a wide arsenal of educational, physiological and manual methods for preventing and treating various health problems, diseases or injuries. In Physiotherapy science, movement is seen as the basis for the individual's total function and as a mean in achieving his goals in relation to the environment. Thus, the individual can affect health through adequate movement and awareness of the body (1). Grotell (2) describes that human movement is a core concept in physical therapy that can continue to be developed both as a practical concept and as a research concept to broaden and deepen the understanding of the complex reality of physical therapy.

Often, individuals' patterns of movement change after injury or illness. The role of the physiotherapist is to support the individual/patient to find a new way or to find a functioning way to move after injury or illness. There are various methods for assessing and analyzing how an individual/patient moves in everyday life and in sports.

One systematic concept for analyzing motion and promoting the basics of effective motion is Joanne Elphinston Movement Systems, JEMSⓇ (3). With the help of structured and severely increased movements, a performance can be improved and developed, which is important both in everyday activities and in sports. The present study is expected to provide knowledge of physiotherapists' experiences and clinical experiences working with the JEMS method in primary care. The study will be conducted as a focus group study.

It is of interest to take note of how the informants reason about concepts such as movement and movement analysis, communication, learning and performance development in the rehabilitation process. By exchanging experiences new knowledge can be formed and the main perspective of the study is expected to shed light on this. The new knowledge can be used in reflection and guidance contexts discussing central concepts. It can also guide the choice of method for motion analysis, treatment and training when implementing rehabilitation methods.

In organisations where time and financial resources are limited, it is important that assessment instruments and treatment methods measure and treat what is useful to most patients. From a socio-economic perspective, it is also important that the patient is offered the right care at the right level of care. The results may constitute a puzzle piece if the method JEMS is perceived by the informants to be an appropriate method to use in primary care for motion analysis and rehabilitation. The results can also be compared with studies on other methods in physiotherapy. Examination of examination and treatment methods is of utmost importance in the selection and implementation of methods in clinical rehabilitation activities.

Physiotherapists are clearly involved in the interprofessional public health work. Early efforts can promote health and improve the functioning of the individual and thus contribute to cost-effectiveness at both individual, business and social levels. Therefore, there is a continuing need for research in physiotherapy and the profession's health promotion, treatment and rehabilitation interventions.

ELIGIBILITY:
Inclusion Criteria:

* the Physiotherapist (PT) has passed the A.R.T courses in JEMS
* the PT is using JEMS in clinical rehabilitation situations on more or less daily bases
* the PT is working in primary care in Region Västra Götaland with employment in public or private care system.

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physiotherapists, male and female, working in primary care in Region Västra Götaland with employment in public or private care system.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
How is it to Work With JEMS: Physiotherapists' Experiences in Working With JEMS, in Primary Care Rehabilitation | 60 to 90 minutes
  The prevalence of Physiotherapists' experiences using the rehabilitation modality JEMS. A focus group study

CONTACTS AND LOCATIONS:
Overall Officials: Jarl, Principal Investigator — Närhälsan Västra Götaland Sweden
Locations (1):
- Monica Johansson, Sollebrunn, Västra Götaland County, Sweden